CLINICAL TRIAL: NCT03033095
Title: Prediction of the Answer to the Treatment by Biotherapies for Naive Spondyloarthritis Disease During 6 Months by Combinatorial Analysis of Serum Biomarkers
Brief Title: Prediction of the Answer to the Treatment by Biotherapies for Naive Spondyloarthritis by Combinatorial Analysis of Serum Biomarkers
Acronym: PRESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 38RC16.018
Record Dates: First submitted 2016-05-11; First posted 2017-01-26 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Spondylitis, Ankylosing
Keywords: TNF inhibitor; Etanercept; Spondyloarthritis; Biomarkers analysis; Personnalized medicine
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- etanercept (Experimental): The etanercept is not the experimental study drug. Etanercept is a treatment justifying the inclusion of patients and is used in accordance with its marketing authorization.
  Modality of administration :
  Etanercept : 50 mg / week subcutaneously, every 7 days The clinical response will be evaluated after 6 months of etanercept treatment, at the M6 visit.
  Interventions: Drug: Etanercept ® 50 mg

INTERVENTIONS:
Drug: Etanercept ® 50 mg — The etanercept is not the experimental study drug. Etanercept is a treatment justifying the inclusion of patients and is used in accordance with its marketing authorization.
  Other Names: ENBREL

SUMMARY:
The aim of this trial is the caracterisation of a predicting algorithm of the answering response for patients with etanercept treatment in spondyloarthritis disease.

This algorithm will help to target patients patients who have a risk / benefit important for etanercept treatment.

DETAILED DESCRIPTION:
Spondyloarthritis (or spondyloarthropathy) is an inflammatory rheumatic disease that causes arthritis. It differs from other types of arthritis because it involves the sites where ligaments and tendons are attached to bones called "entheses."

All patients should get physical therapy and make exercises for joints. Exercises that promote spinal extension and mobility are the most recommended.

Non-steroidal anti-inflammatory drugs (NSAIDs) are the first line treatment for spondylarthritis. NSAIDs are effective when they are used continuously or at the request, in a short or long-term use. However, physicians have to be aware of potential cardiovascular, renal or gastro-intestinal secondary effects when they prescribe NSAIDs. After NSAIDs failure, TNF inhibitors can be used, like infliximab or etanercept. Before starting an anti-TNF treatment, a screening is mandatory. Indeed, patients treated with an anti-TNF must be followed regularly. Until now, there is no algorithm which can predict the response to TNF-inhibitors, and more especially for etanercept treatment.

In this clinical trial, the investigators want to caracterise an algorithm which can predict the response to etanercept for a cohort of patients who suffer from spondyloarthritis.

The development of a predictive algorithm for etanercept treatment will be set up from biological data and finalized with the availibility of clinical data (M6) of the patients .

A modelling by logistic regression will be used, incorporing the set of available variables.

In this clinical trial, the investigators want to caracterise an algorithm which can predict the response to TNF-inhibitors for a cohort of patients with Spondyloarthritis and for an indicated treatment of etanercept.

ELIGIBILITY:
Inclusion Criteria:

* patients with spondylarthritis validating ASAS or New York modified critera, and for who etanercept is indicated.
* Naïve from biological Drug Modifying Anti Rheumatic Drugs
* patients between 18 and 70 years old
* patients who can be monitored at 6 months ;
* patients who can observe the entire treatment ;
* patiens with age to procreate under effective contraception ((abstinence, oral contraceptives , intrauterine devices , implants, spermicide or surgical sterilization ) during the study and for 6 months, 3 weeks after the last injection.
* patients able to understand and accept the terms of the study
* patients having signed the informed consent.
* patients insured under social security

Exclusion Criteria:

* patients of age protected ;
* patients with difficulties for understanding french language ;
* patients with high function disorders incompatible with an education program (dementia Alzheimer's type , etc ...) ;
* patients with psycho- social instability incompatible with regular monitoring (homeless , addictive behavior ,etc.) ;
* patients in a socio- professional situation incompatible with optimal attendance to the program - - Pregnant or nursing patients
* patients who received previously a biotherapy treatment . There is no other exclusion criteria taking into account previous treatments and the duration of them.
* contraindication to the use of anti- TNF treatment
* Surgery scheduled during the study.
* Persons mentioned in Articles L.1121-5 to L.1121-8 of the Public Health Code

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Measurement of disease activity with AS- DAS score (Ankylosing Spondylitis - Disease Activity Score ) | 6 months after inclusion
  An important clinical ASAS response, corresponds to a variation of the ASDAS CRP ≥ 1.1

SECONDARY OUTCOMES:
Measurement of BASDAI response | 6 months after inclusion
  Sensitivity and specificity of the algorithm for BASDAI response : BASDAI response 50, that means an improvement of BASDAI response of 50% or more
biomarkers analysis for personalized medicine | at the inclusion and 6 months after
  8 biomarkers will be analysed :
  * calcium-binding protein complex S100A8/A9,
  * prealbumin,
  * haptoglobin (Hapto),
  * protéine C-réactive (CRP),
  * α1 anti-trypsin
  * apolipoprotéinA1 (ApoA1),
  * platelet factor 4 (PF4),
  * S100A12 protein,

CONTACTS AND LOCATIONS:
Overall Officials: Athan BAILLET, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaltonen KJ, Virkki LM, Malmivaara A, Konttinen YT, Nordstrom DC, Blom M. Systematic review and meta-analysis of the efficacy and safety of existing TNF blocking agents in treatment of rheumatoid arthritis. PLoS One. 2012;7(1):e30275. doi: 10.1371/journal.pone.0030275. Epub 2012 Jan 17. PMID 22272322
- [Background] Braun J, Sieper J. Biological therapies in the spondyloarthritides--the current state. Rheumatology (Oxford). 2004 Sep;43(9):1072-84. doi: 10.1093/rheumatology/keh205. Epub 2004 Jun 8. PMID 15187239
- [Background] Kristensen LE, Saxne T, Nilsson JA, Geborek P. Impact of concomitant DMARD therapy on adherence to treatment with etanercept and infliximab in rheumatoid arthritis. Results from a six-year observational study in southern Sweden. Arthritis Res Ther. 2006;8(6):R174. doi: 10.1186/ar2084. PMID 17121678